CLINICAL TRIAL: NCT06602804
Title: In Vivo 24-Hour Recovery Study of Leukoreduced RBCs Collected on the Trima Accel System Using Non-DEHP Disposable Sets and Stored for 42 Days
Brief Title: Trima Non-DEHP Leukoreduced Red Blood Cell In Vivo Recovery Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCT (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTS-5091
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Device Validation of In-vivo Performance
Keywords: Trima; Trima Accel System; Trima Non-DEHP Disposable Sets; Non-DEHP Disposable Sets; di(2-ethylhexyl) phthalate; Non-DEHP; Red Blood Cell; RBC; Auto RBC; 24-hour red blood cell recovery; Investigational Non-DEHP Disposable Tubing Sets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Healthy adult participants (Experimental): Performance criteria will be evaluated in healthy adult participants, who receive radiolabeled, autologous infusions of LR-RBC components after being stored for 42 days at 2-6°C.
  Interventions: Device: Trima Accel Auto RBC Collection

INTERVENTIONS:
Device: Trima Accel Auto RBC Collection — This is a non-interventional study, observing the in vivo performance of LR-RBC units derived from Trima Accel Auto RBC collection.

SUMMARY:
This is an in vivo 24-hour in-vivo recovery study of leukoreduced red blood cells (RBCs) collected on the Trima Accel System using Non-DEHP disposable sets and stored for 42 days.

ELIGIBILITY:
Inclusion Criteria:

1. Given written informed consent.
2. Age 18 years or older.
3. Normal health status as per AABB criteria for healthy donor.
4. Able to commit to the study schedule.
5. Meets the inclusion criteria defined by site SOPs for automated blood component collection systems or whole blood donation. These criteria are based on AABB standards and FDA regulations.

   a. Note: Participants who are deferred from volunteer community donations due to certain restrictions may participate in the study, as products are not used for allogeneic transfusion; however, sites may or may not implement this depending on their standard procedures.
6. Participants of childbearing potential (either male or female) must agree to use a medically acceptable method of contraception throughout the study.
7. Female participants of childbearing potential must agree to take a pregnancy test prior to the apheresis procedure and prior to reinfusion of radiolabeled LR-RBCs.
8. Participants must agree to report AEs throughout their participation in the study

Exclusion Criteria:

1. Currently pregnant or nursing females.
2. Serum ferritin less than12 ng/mL
3. Has previously completed this study with data included in the EAS.
4. Participation currently, or within the past 30 days, in another investigational trial that would potentially interfere with the analysis of this investigation (eg, pharmaceutical trial).
5. As determined by the Investigator:

   1. Has been diagnosed with a blood disorder(s) affecting RBC characteristics (eg, Glucose 6 Phosphate Dehydrogenase Deficiency [G6PD]),
   2. Reported history of RBC autoantibodies/autoimmune hemolytic anemia, RBC alloantibodies,
   3. Clinically significant acute or chronic disease, or
   4. Reported history of hypersensitivity to technetium or chromium
   5. Other unspecified reason that, in the opinion of the Investigator, makes the healthy adult volunteer unsuitable for enrollment.
6. Treatment with any medication as specified in site deferral list (based on AABB medication deferral list for apheresis donors).
7. Previously transfused/reinfused with RBCs within the last 120 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-08-26 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Success of RBCs in Vivo Recovery After 42-day Storage | 43 days
  The primary outcome of this study is to demonstrate that LR-RBCs collected on the Trima Accel system using non-DEHP disposable tubing sets with AS-3 meet the FDA criteria for 24-hour recovery after 42 days of refrigerated storage in non-DEHP storage bags.
  The 3 parts of FDA RBC recovery criteria that must be met (below) are presented in Primary Outcome 1 and Primary Outcome 2. The derivation of the sample size was based on the level of precision attained with 26 subjects relative to the 1st part of the criteria.
  1. A one-sided lower confidence limit for the proportion of RBC components with 24-hour RBC in vivo recovery less than 75% is 70%* (Primary Outcome 1),
     *Allows for low recoveries (greater than 75%) in up to 3 out of 24 to 26 participants
  2. A sample mean of in vivo 24-hour RBC percent recovery ≥ 75% (Primary Outcome 1)
  3. A sample standard deviation of in vivo 24-hour percent RBC recovery ≤ 9% (Primary Outcome 2)
Mean 24-hour, Post-transfusion, In Vivo RBC Recovery Percentage After 42-day Storage | 43 days
  The primary outcome of this study is to demonstrate that LR-RBCs collected on the Trima Accel system using non-DEHP disposable tubing sets with AS-3 meet the FDA criteria for 24-hour recovery after 42 days of refrigerated storage in non-DEHP storage bags.
  The 3 parts of FDA RBC recovery criteria that must be met (below) are presented in Primary Outcome 1 and Primary Outcome 2. The derivation of the sample size was based on the level of precision attained with 26 subjects relative to the 1st part of the criteria.
  1. A one-sided lower confidence limit for the proportion of RBC components with 24-hour RBC in vivo recovery less than 75% is 70%* (Primary Outcome 1),
     *Allows for low recoveries (greater than 75%) in up to 3 out of 24 to 26 participants
  2. A sample mean of in vivo 24-hour RBC percent recovery ≥ 75% (Primary Outcome 1)
  3. A sample standard deviation of in vivo 24-hour percent RBC recovery ≤ 9% (Primary Outcome 2)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Hoxworth Blood Center, University of Cincinnati College of Medicine, Cincinnati, Ohio
  - American Red Cross, Norfolk Clinical Research Lab, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No
Privacy concerns